CLINICAL TRIAL: NCT04996550
Title: Cluster and Registry Trial of the Working Group of Heart Failure in Denmark. Are Carvedilol and Metoprolol Succinate Comparable Treatments in Heart Failure Patients With Reduced Ejection Fraction
Brief Title: Are Carvedilol and Metoprolol Succinate Comparable Treatments in Heart Failure Patients With Reduced Ejection Fraction
Acronym: CROWD-COMPARE
Status: Not yet recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mikael Kjaer Poulsen, Principal Investigator, Odense University Hospital
Other Study IDs: CROWD-COMPARE
Record Dates: First submitted 2021-07-29; First posted 2021-08-09 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Chronic Heart Failure
MeSH Terms: interventions — Carvedilol; Metoprolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Carvedilol group: Treated with Carvedilol
  Interventions: Drug: Carvedilol
- Metoprolol succinate group: Treated with Metoprolol succinate
  Interventions: Drug: Metoprolol Succinate

INTERVENTIONS:
Drug: Carvedilol — To compare the efficacy of carvedilol and metoprolol succinate on all-cause mortality or first hospitalization for worsening heart failure in patients with heart failure with reduced ejection fraction with an indication for treatment with beta-blockers.
  Groups: Carvedilol group
Drug: Metoprolol Succinate — To compare the efficacy of carvedilol and metoprolol succinate on all-cause mortality or first hospitalization for worsening heart failure in patients with heart failure with reduced ejection fraction with an indication for treatment with beta-blockers.
  Groups: Metoprolol succinate group

SUMMARY:
The objective of CROWD-COMPARE is to compare the efficacy of carvedilol and metoprolol succinate on all-cause mortality or first hospitalization for worsening heart failure in patients with heart failure with reduced ejection fraction with an indication for treatment with beta-blockers.

DETAILED DESCRIPTION:
Background:

Heart failure with reduced ejection fraction:

The overall prevalence of heart failure with reduced ejection fraction (HFrEF) is 1-2% in the adult population and increasing with age to more than 10% in the population over 70 years. Patients with HFrEF have markedly reduced life expectancy, physical capacity and quality of life. Activation of the sympathetic nervous system is one of the cardinal pathophysiologic abnormalities in patients with HFrEF. Levels of circulating catecholamines increase in patients with HFrEF in proportion to the severity of the disease and those with the highest plasma levels of norepinephrine have the most unfavorable prognosis.

Beta-blocker in heart failure with reduced ejection fraction:

Prospective randomized clinical trials of sympathetic antagonists with several different beta-blockers have shown that these medications can reduce symptoms, improve left ventricular function, increase functional capacity, decrease the number of hospitalization for worsening heart failure and mortality in patients with HFrEF. Current heart failure guidelines therefore recommend treatment with a beta-blocker in HFrEF patients as a class 1A indication. However, small differences exist between beta-blockers. Metoprolol is a second generation beta-blocker that selectively inhibit β1-adrenoceptors, whereas carvedilol is a third generation beta-blocker, that nonselectively inhibit β1-adrenoceptors with additional inhibition of α1-adrenoceptors. Therefore, controversy exists whether beta-blockers exert a class effect or whether one beta-blocker is superior to another. In the largest prospective randomized clinical trial that directly compared the efficacy of beta-blockers, the Carvedilol or Metoprolol European Trial (COMET), carvedilol increased survival in patients with HFrEF compared with metoprolol tartrate. However, the results of the COMET trial was debated for two reasons. First, it compared carvedilol with the short-acting metoprolol tartrate formulation. Metoprolol tartrate, however, is not the formulation used in key HFrEF metoprolol trials and is not recommended in current heart failure guidelines. Second, the metoprolol tartrate target dose in the COMET trial was 50 mg twice daily, whereas the long-acting metoprolol succinate dose in the Metoprolol CR/XL Randomized Intervention Trial (MERIT) trial was 200 mg once daily,10 as recommended by the heart failure guidelines. Further, Carvedilol was dosed at full guideline target dose in COMET.

No pharmaceutical company has shown interest in carrying out such a comparative study. Attempts have been made to compare these medications based on information from different studies, but these so-called network meta-analyses are severely hampered by having different inclusion and exclusion criteria, different end-points, ect. At the same time the patent of both carvedilol and metoprolol succinate has expired in Denmark.

Objectives:

The objective of CROWD-COMPARE is to compare the efficacy of carvedilol and metoprolol succinate on all-cause mortality or first hospitalization for worsening heart failure in patients with heart failure with reduced ejection fraction with an indication for treatment with beta-blockers.

Methods:

Design and cluster allocation:

CROWD-COMPARE is a crossover comparative effectiveness study with random allocation of clusters. Each participating department of cardiology will be allocated to four periods (clusters): two periods with carvedilol as the principal beta-blocker and two periods with metoprolol succinate as principal beta-blocker. Departments will be randomly allocated as to whether they will begin with the carvedilol or the metoprolol succinate cluster and then alternate between clusters annually.

If a cluster becomes scheduled to stop before four years due to organizational changes (eg. if the department of cardiology associated heart failure clinic is closed or merged with another clinic), the investigators may change the duration of the remaining periods for that cluster in order to get compatible allocation periods for the two medications.

Eligible departments:

All 23 danish departments of cardiology with a heart failure clinic associated, which report to the Danish Heart Failure Registry are eligible.

Treatment in allocation arms:

Treatment in clusters will adhere to Danish and European guidelines, where the indication for beta-blocker treatment is symptomatic heart failure (NYHA ≥ II) with LVEF ≤40%. There is no difference in indication or contraindications for the two medications. Carvedilol or metoprolol succinate will be titrated to target dose (Carvedilol 25 mg twice daily or metoprolol succinate 200 mg once daily) or the maximal tolerated dose according to standard heart failure care. There will not be any extra patient visits due to the study.

Data collection during the allocation period:

As the respective departments of cardiology with an associated heart failure clinic are cluster randomized, there will be no study-related collection of data on individual patients during the allocation period. All data will be obtained from national registries.

Follow-up:

For the purpose of follow-up, data from the Danish Heart Failure Registry, which is routinely uploaded to Statistics Denmark, will be linked in anonymous form to hospital admissions, diagnosis, vital status, cause of death, dispensed descriptions and biochemistry from The Danish National Patient Registry, The Danish Civil Registration System, The Clinical Laboratory Information System and the Danish National Prescription Registry.

The National Prescription Registry entries in Statistics Denmark have a delay of 12 to 18 months, while vital status and admissions are updated with only a few months delay. Hence, the primary endpoint will be assessed two years after the end of the 4-year allocation period. At that time, we will be able to identify patients, who have filled in a prescription for carvedilol or metoprolol succinate during the allocation period. Further, we will have data on survival and hospital admission for a minimum follow-up period of two years.

Data management plan:

All data will be stored and analyzed on the Statistics Denmark servers through our agreement with the Division of Research Services at Statistics Denmark. There is no extra storage of data in relation to this scientific study.

Analysis:

Primary endpoint:

The primary endpoint will be a combined endpoint of all-cause mortality or first hospitalization for worsening heart failure. To have adequate statistical power, we will need an overall event rate of 15% (840 events) for the primary outcome.

Primary analysis:

Proportional hazard regression of time to the primary endpoint from time of first claiming a prescription for carvedilol or metoprolol succinate, comparing carvedilol clusters with metoprolol succinate clusters adjusted for department of cardiology.

Secondary endpoints

* All-cause mortality
* A combined endpoint of all-cause mortality or first hospitalization for worsening heart failure according to heart rhythm (sinus rhythm or atrial fibrillation/flutter)

Secondary analyses:

* Cost-effectiveness analysis of each strategy
* Proportion of patients who remained on beta-blocker treatment for a minimum of one year
* Proportion of patients who switched from their initially prescribed beta-blocker to the other
* Proportion of patients who reached target dose

Intention to treat cohort:

Analyses will be performed on all participating departments of cardiology with an associated heart failure clinic, which report data to the Danish Heart Failure Registry during the study period.

Sample size considerations:

Based on data from the Danish Heart Failure Registry, we expect that 2700 patients annually will be candidates for the treatment with either carvedilol or metoprolol succinate. Some of these patients will already be on betablockers before first visit or hospitalization. In the Danish Heart Failure Registry, 1-year mortality is 10%. With 23 clusters and an estimated overall rate of the primary endpoint of 15% (see above for description of primary endpoint), we will need to recruit registry data from 1400 patients per year (5600 patients in total) to obtain 840 events over a period of four years to detect at relative reduction of 20% between treatment groups with a significance level of 5% and a power of 90% (α=0.05, β=0.10).

Statistics:

Analyses will be performed according to the CONSORT statement recommendation for cluster trials. Statistical analyses will be performed using commercially or open-source available statistical software. Primary results will be assessed as intention-to-treat. In addition, we will conduct an instrumental variable analysis, where the cluster randomization is used as an instrument for actually received treatment. In case of low-compliance to the cluster allocated treatment then instrumental variables is the only way to estimate the causal effect. Continuous data will be presented as median (25-75% range). A two-tailed p value of 0.05 or less is considered statistically significant.

Results for subgroups will be presented. These will be prespecified prior to trial termination.

Ethical aspects:

The two beta-blockers are considered equal in Danish and European heart failure guidelines. Participating departments of cardiology will continue to follow best practice, with each department having one of the two beta-blockers as principal option at a given period of time. Departments who do not wish to switch between principal beta-blockers will not be included. Of importance, all patients will be prescribed the medication that is considered best for them. Hence, all patients will receive the same individually tailored treatment as patients do today at their respective department of cardiology.

Patients will be informed about the trial in two ways: 1) by a posted bulletin in the department stating that the department is participating in CROWD-COMPARE, and 2) by the treating physician informing them, upon prescribing the beta-blocker, that the department is participating in a national effort to compare two equivalent medications, which according to heart failure guidelines are both first-line choices, and that currently the department of cardiology is using the prescribed medication in cases where the patient and treating physician after individual assessment do not have a preference for either beta-blocker.

The price difference between the two beta-blockers varies, but is less than 0.50,- kr./day. (Daily cost: carvedilol 25 mg x 2: 0.63,- kr./day. versus metoprolol succinate 200 mg x 1: 0.57,- kr./day. (April the 30th, 2021). For this reason, the current study will not cause the individual patient nor society (as the patient receives state sponsored premiums for their medications) substantial extra expenses. In case of side effects after the initiation of a beta-blocker, patients can be changed to the other at the discretion of the clinician. The study does not result in extra visits for the patients.

The study follows the Helsinki Declaration II.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* NYHA ≥ II
* LVEF ≤40%

Exclusion Criteria:

* No indication for beta-blocker treatment or contraindications for the two for the two study drugs (Carvedilol or metoprolol succinate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All 23 danish departments of cardiology with a heart failure clinic associated, which report to the Danish Heart Failure Registry are eligible.
Sampling Method: Probability Sample
Enrollment: 5600 (Estimated)
Dates: Start 2022-01-03 (Estimated); Primary Completion 2028-01-02 (Estimated); Study Completion 2028-12-18 (Estimated)

PRIMARY OUTCOMES:
A combined endpoint of all-cause mortality or first hospitalization for worsening heart failure. | Four years with randomized cluster allocation and two year of follow-up.
  To compare the efficacy of carvedilol and metoprolol succinate in patients with heart failure with reduced ejection fraction with an indication for treatment with beta-blockers.

SECONDARY OUTCOMES:
All-cause mortality. | Four years with randomized cluster allocation and two year of follow-up.
  To compare the efficacy of carvedilol and metoprolol succinate in patients with heart failure with reduced ejection fraction with an indication for treatment with beta-blockers.
A combined endpoint of all-cause mortality and first hospitalization for worsening heart failure according to heart rhythm (sinus rhythm or atrial fibrillation/flutter). | Four years with randomized cluster allocation and two year of follow-up.
  To compare the efficacy of carvedilol and metoprolol succinate in patients with heart failure with reduced ejection fraction with an indication for treatment with beta-blockers.

OTHER OUTCOMES:
Cost-effectiveness analysis of each strategy. | Four years with randomized cluster allocation and two year of follow-up.
  To compare the efficacy of carvedilol and metoprolol succinate in patients with heart failure with reduced ejection fraction with an indication for treatment with beta-blockers.
Proportion of patients who remained on beta-blocker treatment for a minimum of one year. | Four years with randomized cluster allocation and two year of follow-up.
  To compare the efficacy of carvedilol and metoprolol succinate in patients with heart failure with reduced ejection fraction with an indication for treatment with beta-blockers.
Proportion of patients who switched from their initially prescribed beta-blocker to the other. | Four years with randomized cluster allocation and two year of follow-up.
  To compare the efficacy of carvedilol and metoprolol succinate in patients with heart failure with reduced ejection fraction with an indication for treatment with beta-blockers.
Proportion of patients who reached target dose. | Four years with randomized cluster allocation and two year of follow-up.
  To compare the efficacy of carvedilol and metoprolol succinate in patients with heart failure with reduced ejection fraction with an indication for treatment with beta-blockers.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Odense University Hospital, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No
Final results.